CLINICAL TRIAL: NCT05885932
Title: Drug-eluting Stenting Versus Medical Treatment Alone for Patients With Extracranial Vertebral Artery Stenosis: The VISTA Trial
Brief Title: Drug-eluting Stenting Versus Medical Treatment for Extracranial Vertebral Artery Stenosis
Acronym: VISTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VISTA
Record Dates: First submitted 2023-05-07; First posted 2023-06-02 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-05

CONDITIONS: Ischemic Stroke; Vertebral Artery Stenosis
Keywords: Extracranial vertebral artery stenosis; Drug-eluting stenting; Best medical treatment; Ischemic stroke
MeSH Terms: conditions — Ischemic Stroke; Vertebrobasilar Insufficiency | interventions — Aspirin; Clopidogrel; Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-eluting stenting group (Experimental): All the participants in this group will be performed with extracranial vertebral artery sirolimus-eluting stenting plus best medical treatment including Aspirin 100mg per day + Clopidogrel 75mg per day or Ticagrelor 90mg twice per day for 6 months and mono anti-platelet therapy thereafter.
  Interventions: Procedure: Drug-eluting stenting plus aspirin and clopidogrel or ticagrelor
- Medical group (Active Comparator): All the participants in this group will be given medical therapy including Aspirin 100mg per day + Clopidogrel 75mg per day or Ticagrelor 90mg twice per day for 6 months and mono anti-platelet therapy thereafter.
  Interventions: Drug: Aspirin and clopidogrel or ticagrelor; Procedure: mono anti-platelet therapy

INTERVENTIONS:
Procedure: Drug-eluting stenting plus aspirin and clopidogrel or ticagrelor — All the participants in this group will be performed with extracranial vertebral artery sirolimus-eluting stenting plus medical therapy including aspirin 100mg per day + clopidogrel 75mg per day or ticagrelor 90mg twice per day for 6 months and mono anti-platelet therapy thereafter.
  Other Names: Sirolimus-eluting stenting plus dual antiplatelet therapy
  Arms: Drug-eluting stenting group
Drug: Aspirin and clopidogrel or ticagrelor — All the participants in this group will be given medical therapy including aspirin 100mg per day + clopidogrel 75mg per day or ticagrelor 90mg twice per day for 6 months and mono anti-platelet therapy thereafter.
  Arms: Medical group
Procedure: mono anti-platelet therapy — mono anti-platelet therapy
  Arms: Medical group

SUMMARY:
Posterior circulation stroke accounts for 20% of all ischemic stroke. Approximately one quarter of posterior circulation strokes are due to stenosis in the vertebral artery and basilar artery.

Two previous randomized controlled trials focusing on vertebral artery stenting, the Vertebral Artery Stenting Trial (VAST) and the Vertebral Artery Ischaemia Stenting Trial (VIST) were underpowered because they failed to reach target recruitment, and both the trials found no difference in risk of the primary outcome between the stenting group and medical group.

The drug-eluting stenting versus medical therapy alone for patients with extracranial vertebral artery stenosis (VISTA) trial, is a government-funded, prospective, multicenter, randomized controlled trial. It will recruit patients with 3 months stroke or TIA caused by 70-99% stenosis of extracranial vertebral artery (V1-2 segments). Only high-volume center with a proven track record will enroll patients. Patients will be randomized (1:1) to best medical treatment alone or medical treatment plus stenting. Primary outcome is a composite of any fatal or non-fatal stroke within 30 days after randomization, or ischemic stroke in the territory of the target artery beyond 30 days to 1 year. The VISTA trial will be conducted in 30 sites in China and aims to have a sample size of 472 subjects (stenting, 236; medical treatment, 236). Recruitment is expected to be finished by Sep, 2025. Patients will be followed for 1 year at first stage. Long-term follow-ups till 3 years or longer is also preplanned. The first stage of the trial is scheduled to complete in 2027.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Extracranial vertebral artery (V1-2 segments) has 70% to 99% stenosis (NASCET criteria by angiography), and the diameter of the target vessel ≥ 2.5mm.
3. History of clinical symptoms associated with target vessels within 3 months before randomization, including ischemic stroke (modified Rankin Scale, mRS score ≤ 3) or transient ischemic attack (TIA).
4. With more than two atherosclerotic risk factors such as, hypertension, hyperlipidemia, diabetes, smoking, drinking, obesity, or obstructive sleep apnea (following the 2021 AHA/ASA guidelines).
5. mRS score ≤ 3.
6. Patients or their guardians voluntarily participate of the study and sign the consent form.

Exclusion Criteria:

1. Vertebral artery stenosis caused by non-atherosclerotic lesions, including arterial dissection, Moyamoya disease, vasculitis disease, radiation-induced vascular disease, fibromuscular dysplasia, etc.
2. Tandem extracranial or intracranial severe stenosis or occlusion of the target vessel.
3. History of open surgery or endovascular treatment of the target vessel.
4. Other cerebrovascular diseases that require one-stage open surgery or endovascular therapies.
5. Open surgery or endovascular treatment for other cerebrovascular diseases within 1 month.
6. Patients in whom vertebral anatomy was felt to be technically not feasible for vertebral artery stenting (e.g. access problems).
7. The contralateral vertebral artery and basilar artery have lesions that may be related to the symptoms, and the investigators cannot confirm that the target vessel is the responsible vessel for the symptoms (For example, the ostium of bilateral vertebral artery is severely narrowing, and the diameter of vertebral artery is equal, unable to determine the dominant vertebral artery).
8. Known allergy or contraindication to iodinated contrast media and sirolimus.
9. History of acute ischemic stroke within 7 days.
10. History of intracranial hemorrhage, subarachnoid hemorrhage, subdural hemorrhage, or extradural hemorrhage within 6 weeks.
11. Cardioembolic strokes as evident by prior history of strokes in other territories or multi-territory strokes in the presence of risk factors known to be associated with cardiogenic embolism (e.g. atrial fibrillation, left ventricular thrombus or history of myocardial infarction within 6 weeks, etc.).
12. Coagulation dysfunction or hemorrhagic tendency (e.g. INR > 1.5 and/or platelet count < 100×10^9/L).
13. Cannot complete the follow-up due to severe diseases (e.g. serious infections, severe chronic obstructive pulmonary disease, malignancy, dementia, mental illness, uncontrolled server hypertension or diabetes).
14. Women who are pregnant or lactating.
15. According to the judgement of the investigator, other situations, influencing the safety and efficacy evaluation, which make the patient not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 472 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Any fatal or non-fatal stroke within 30 days after randomization, or ischemic stroke in the territory of the target artery beyond 30 days to 1 year. | 1 year
  The number of participants who suffer from any fatal or non-fatal stroke within 30 days after randomization, or ischemic stroke in the territory of the target artery beyond 30 days to 1 year.

SECONDARY OUTCOMES:
Fatal or non-fatal stroke within 30 days | within 30 days
  The number of participants who suffer from fatal or non-fatal stroke within 30 days after randomization.
Ischemic stroke in the territory of the target artery beyond 30 days to 1 year | beyond 30 days to 1 year
  The number of participants who suffer from ischemic stroke in the territory of the target artery beyond 30 days to 1 year.
Ischemic stroke in the territory of the target artery within 1 year | within 1 year
  The number of participants who suffer from ischemic stroke in the territory of the target artery within 1 year.
Crescendo TIA in the territory of the target artery within 1 year | within 1 year
  The number of participants who suffer from crescendo TIA in the territory of the target artery within 1 year.
Fatal stroke within 1 year | within 1 year
  The number of participants who suffer from fatal stroke within 1 year.
Disabling stroke (defined by a modified Rankin Scale Score of ≥3) within 1 year | within 1 year
  The number of participants who suffer from disabling stroke (defined by a modified Rankin Scale Score of ≥3) within 1 year.
Any stroke within 1 year | within 1 year
  The number of participants who suffer from any stroke within 1 year.
Any stroke, myocardial infarction or death within 1 year | within 1 year
  The number of participants who suffer from any stroke, myocardial infarction or death within 1 year.
All cause mortality within 1 year | within 1 year
  The number of participants who die of any cause within 1 year.
Symptomatic cerebral hemorrhage within 1 year | within 1 year
  The number of participants who suffer from symptomatic cerebral hemorrhage within 1 year.
Modified Rankin Scale (mRS) score (0-5, higher score refers to a worse outcome) | at 1 year
  Modified Rankin Scale (mRS) score at 1 year.
In-stent restenosis (Stenosis ≥ 50%) | at 1 year
  In-stent restenosis (Stenosis ≥ 50%) at 1 year. Performing CTA or DSA to evaluate the stenosis degree.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University., Beijing, China

IPD SHARING:
Plan to Share IPD: No